CLINICAL TRIAL: NCT05191238
Title: Patients Pull the Strings: A Pilot Study of IUD Self-Removal Simulation
Brief Title: Intrauterine Device (IUD) Self Removal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of difficulty recruiting participants.
Sponsor: Boston Medical Center (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-42042
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: IUD Removal
Keywords: Self removal of IUD; Educational video; Simulation; Patient education; Intrauterine device; Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants consented for IUD removal (Experimental): Participants will be shown an educational video about IUD self-removal and simulation models. After the video, participants will be given the choice to either attempt IUD self-removal or to have their provider perform standard removal. If a participant elects to attempt self-removal and fails, their provider will offer standard removal.
  Interventions: Other: IUD self-removal education

INTERVENTIONS:
Other: IUD self-removal education — Two part educational intervention (watching IUD self-removal video and practicing IUD removal on two simulation models)

SUMMARY:
This pilot research study will teach patients how to self-remove intrauterine contraceptive device (IUD) through an educational video and simulation and evaluate patient perspectives and experiences related to IUD self-removal with two surveys. Patients will be recruited for this study at the time of presentation to the office for IUD removal. After consenting to the procedure, participants will complete a pre-intervention survey, watch a video explaining how to self-remove the IUD, and use two models to simulate IUD removal. After completion of using the models to practice IUD removal, participants will complete a second short survey. The participant will then be given the option of attempting self-removal and be given time to attempt the removal. If the participant elects to have the provider remove their IUD, the provider will do so. At the end of the encounter, participants will fill out a final survey. Research staff will measure the length of the strings of all IUDs prior to routine disposal of the device.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Present to Boston Medical Center Yawkey for removal of IUD and have been consented for removal
* Are eligible for removal of IUD in the office setting

Exclusion Criteria:

* Current incarceration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Change in proportion of participants who are willing to attempt IUD self-removal | baseline, 15-30 minutes
  Participants will be asked before and after reviewing the educational video and practicing self-removal through simulation, if they are willing to attempt IUD self-removal. The change in the proportion willing to attempt IUD self-removal will be calculated.
Proportion of participants who attempt IUD self-removal | 15-30 minutes
  Attempt Yes/No

SECONDARY OUTCOMES:
Success of IUD self removal | 1 day
  Success Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Wong, MD, Principal Investigator — Boston Medical Center, Obstetrics and Gynecology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No